CLINICAL TRIAL: NCT06379243
Title: Development and Validation of a Postoperative Re-fracture Risk Model for Osteoporotic Spinal Fractures: a Multicenter Prospective Cohort Study
Brief Title: Development and Validation of a Postoperative Re-fracture Risk Model for Osteoporotic Spinal Fractures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Seventh Affiliated Hospital of Sun Yat-sen University (Other)
Collaborators: Guangzhou Medical University (Other); Huizhou Municipal Central Hospital (Other); Dongguan Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Qingyu Liu, chief physician, The Seventh Affiliated Hospital of Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KY-2023-008-02
Record Dates: First submitted 2024-04-17; First posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Osteoporosis Fracture; Osteoporosis Vertebral; Compression Fracture; Perform PVP / PKP Treatment
Keywords: osteoporosis; spinal vertebral fractures; PVP / PKP treatment
MeSH Terms: conditions — Osteoporotic Fractures; Fractures, Compression; Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- non-operative vertebra refracture (Experimental): observe non-operative vertebra refracture after PVP/PKP surgery.
  Interventions: Procedure: PVP/PKP

INTERVENTIONS:
Procedure: PVP/PKP — PVP or PKP surgery in patients with osteoporotic vertebral compression fractures

SUMMARY:
In this project, IDEAL-IQ technology and PDFF and R2* image-based imaging methods are used to analyze the intrinsic relationship between preoperative vertebral bone marrow fat content, magnetic susceptibility properties of bone tissue and bone strength (bone volume and bone mass), to explore the mechanism of vertebral re-fracture after PVP / PKP, and to explore the imaging markers for the risk of postoperative vertebral re-fracture after PVP / PKP. To construct a precise and individualized risk assessment model of vertebral re-fracture after PVP/ PKP by combining clinical risk factors, preoperative quantitative MRI parameters (PDFF, R2*) and imaging characteristics, so as to achieve the goal of objectively and accurately evaluating the risk of vertebral re-fracture at the early stage of the postoperative period (1 year).

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with osteoporotic vertebral fractures of the thoracic and lumbar level with reference to the 2022 edition of the Osteoporotic Fractures Guidelines (2022 edition);
* The presence of bone marrow edema or hemorrhage (acute fracture) in the fractured vertebrae is clearly defined by MR examination, and the responsible vertebrae is treated with PVP / PKP;
* Number of fractured vertebrae: 1-3 vertebral compression fractures (including old fractures).

Exclusion Criteria:

* History of severe scoliosis, vertebroplasty, or internal spinal fixation;
* Presence of spinal infection and malignant neoplastic disease;
* Presence of mental disease, cognitive impairment, or critical illness (e.g., severe cardiac or cerebrovascular disease).

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Non-operative vertebral re-fracture within 1 year after PVP / PKP | 1 year
  Non-operative vertebral re-fracture within 1 year after PVP / PKP, confirmed by follow-up spinal MRI

SECONDARY OUTCOMES:
Visual Analog Score (VAS) at 1 year after PVP/ PKP | 1 year
  Visual Analog Score (VAS) at 1 year after PVP / PKP were obtained by completing the appropriate questionnaires on-site at the time of the 1-year postoperative spinal MRI review.
Oswestry Dysfunction Index (ODI) at 1 year after PVP/PKP | 1 year
  Oswestry Dysfunction Index (ODI) at 1 year after PVP / PKP were obtained by completing the appropriate questionnaires on-site at the time of the 1-year postoperative spinal MRI review.

CONTACTS AND LOCATIONS:
Overall Officials: qingyu liu, Principal Investigator — The Seventh Affiliated Hospital of Sun Yat-sen University
Locations (1):
- The Seventh Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No